CLINICAL TRIAL: NCT07330700
Title: "A Single-Blind Randomized Controlled Trial to Investigate the Effects of Marching Exercise Combined With Cognitive Training on Physical Performance, Cognitive Function, and Autonomic Cardiovascular Responses in Older Adults With Type 2 Diabetes Mellitus"
Brief Title: Effects of Marching Exercise With Cognitive Training on Physical, Cognitive Function, and Autonomic Cardiovascular Responses in Older Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonticha Kaewjoho (Other)
Collaborators: University of Phayao (Other)
Responsible Party: Sponsor-Investigator, Chonticha Kaewjoho, Chonticha Kaewjoho, University of Phayao
Organization: University of Phayao (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPhayaoChonticha-221
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Type2 Diabetes Mellitus; Autonomic Nervous System Imbalance
Keywords: Type2 Diabetes Mellitus; Dual-task Exercise; Marching Exercise; Autonomic Nervous System; Heart Rate Variability
MeSH Terms: interventions — MME

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three parallel groups:
  1. Modified Marching Exercise combined with cognitive training
  2. Modified Marching Exercise alone, or
  3. Control group receiving usual care. Outcomes are assessed before and after the 6-week intervention period.
Who Masked: Participant
Masking Description: Participants are blinded to group allocation. Due to the nature of the exercise interventions, care providers and investigators are not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modified Marching Exercise combined with Cognitive Training (Experimental): Participants in this group perform a Modified Marching Exercise combined with dual-task cognitive training. The exercise consists of rhythmic marching movements while simultaneously performing cognitive tasks such as backward counting and reciting months in reverse order. Each session lasts approximately 30 minutes and is conducted according to the assigned intervention protocol.
  Interventions: Other: Modified Marching Exercise combined with cognitive training group
- Modified Marching Exercise (Experimental): Participants in this group perform the Modified Marching Exercise alone without concurrent cognitive tasks. The exercise involves rhythmic marching movements adapted to individual functional ability. Each session lasts approximately 30 minutes and follows the same frequency and duration as the experimental intervention.
  Interventions: Other: Modified Marching Exercise group
- Control group (No Intervention): Participants in the control group receive health education and educational pamphlets focused on fall prevention. They continue their usual daily activities without participation in a structured exercise program during the study period.

INTERVENTIONS:
Other: Modified Marching Exercise combined with cognitive training group — The exercise program consists of a Modified Marching Exercise that emphasizes lifting the knees to touch a designated rope during each step. A metronome is used to maintain a rhythmic pace of 60-80 beats per minute throughout the training.
  In addition, participants perform concurrent cognitive dual-task training designed to stimulate executive function. The cognitive tasks include countdown calculations, backward sequencing of months and weekdays, and a Stroop interference task.
  Each session lasts approximately 30-40 minutes and includes a 5-minute warm-up and a 5-minute cool-down. Exercise intensity is individually adjusted according to the participant's fitness level. The program is conducted three times per week for 6 consecutive weeks, for a total of 18 sessions.
  This combined cognitive-motor training is designed to integrate physical and cognitive demands in order to improve movement efficiency, balance control, and responses to daily functional stimuli.
  Other Names: MME with Dual-task Marching Exercise
  Arms: Modified Marching Exercise combined with Cognitive Training
Other: Modified Marching Exercise group — Participants perform a structured Modified Marching Exercise program. The exercise involves rhythmic marching movements with pace controlled by a metronome set at 80 beats per minute. The intervention is conducted three sessions per week for 6 weeks, with each session lasting approximately 30-40 minutes, including warm-up and cool-down periods. All exercise sessions are supervised by a licensed physical therapist.
  Other Names: MME
  Arms: Modified Marching Exercise

SUMMARY:
This study aims to evaluate the effects of a combined marching exercise with cognitive training program on physical performance, cognitive function, and autonomic cardiovascular responses in older adults with type 2 diabetes mellitus. Participants will be randomly assigned to either an intervention group receiving marching exercise with cognitive tasks or a control group receiving usual care. Outcomes will be assessed before and after the intervention period. The findings are expected to provide evidence for a feasible and safe exercise strategy to improve physical and cardiovascular health in older adults with type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is highly prevalent among older adults and is associated with declines in physical function, cognitive performance, and autonomic cardiovascular regulation. Reduced physical activity and impaired autonomic nervous system function may increase the risk of functional limitation, falls, and cardiovascular complications in this population. Exercise interventions that simultaneously challenge physical and cognitive domains may provide additional benefits beyond conventional exercise alone.

This single-blind, randomized controlled trial investigates the effects of a marching exercise program combined with cognitive training on physical function, cognitive performance, and autonomic cardiovascular responses in older adults with type 2 diabetes mellitus. Eligible participants aged 60 years and older will be recruited from the community and randomly assigned to either an intervention group or a control group.

The intervention group will participate in a structured marching exercise program integrated with cognitive tasks, conducted three times per week for eight weeks. The control group will receive usual care and standard health advice. Physical performance outcomes will include measures of mobility, balance, and cardiorespiratory fitness. Cognitive function will be assessed using standardized cognitive tasks. Autonomic cardiovascular responses will be evaluated using heart rate variability parameters.

Outcome measures will be assessed at baseline and after completion of the intervention. This study aims to provide clinical evidence supporting a practical and community-based dual-task exercise approach for improving physical, cognitive, and autonomic cardiovascular health in older adults with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female.
2. Aged between 60 and 79 years.
3. Medically diagnosed with type 2 diabetes.
4. Peripheral neuropathy with a score of 7 or higher according to the Michigan Neuropathy Screening Instrument (MNSI).
5. Body Mass Index (BMI) within the normal range (between 18.5-24.5 kg/m²).
6. Able to follow instructions and willing to participate in the study.
7. Able to communicate with researchers and provide information independently (researchers will read the questions to the volunteers and allow them to choose their own answers).
8. Able to walk continuously for at least 10 meters without the use of walking aids.

Exclusion Criteria:

1. Neurological disease (e.g., stroke, Parkinson's disease, spinal cord injury) that affects mobility, such as balance and gait.
2. Open wounds on the skin that affect weight-bearing while standing or walking. 1) Deformities or abnormalities of the extremities, or disabilities resulting from the loss of limbs that may affect the study.

2) Inflammation of joints and muscles, or musculoskeletal conditions with a pain score greater than 5 out of 10 on the Visual Analogue Scale (VAS), or any pain that affects the study.

3) A history of ankle, knee, or hip joint replacement within 6 months prior to participation in the study, or any residual effects from surgery that affect the study.

4) Hearing and vision impairments that cannot be corrected with hearing aids and glasses, etc.

5) Other complications that may affect the study, such as dizziness, angina pain, uncontrolled high blood pressure, acute illness, or injury, etc.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | Baseline, immediately after 6 weeks of intervention, and 1-month follow-up
  Heart Rate Variability (HRV) Assessment HRV is assessed using the SA-3000P device to evaluate Autonomic Nervous System (ANS) function, stress resistance, and arterial elasticity. The procedure involves a 3-minute measurement using a finger probe while the subject sits quietly. The device automatically analyzes the data to provide time-domain indices (such as SDNN), which are used to assess cardiac function and prognosis.
Handgrip strength test | Baseline, immediately after 6 weeks of intervention, and 1-month follow-up
  Handgrip Strength Testing This test assesses hand and forearm muscle strength using a hand grip dynamometer. The subject stands upright with the dominant arm extended alongside the body (abducted approx. 15 degrees), elbow straight, and palm facing down. Upon the "start" signal, the subject squeezes the device as hard as possible.
Five times sit-to-stand test (FTSST) | Baseline, immediately after 6 weeks of intervention, and 1-month follow-up
  Leg Muscle Strength Test (FTSST) The Five Times Sit to Stand Test measures leg strength using a standard armless chair. The subject performs five consecutive stand-to-sit cycles as quickly and safely as possible from a seated position (hips ~90°). Time is recorded from the start signal until the final return to sitting. The average of three trials is calculated (Kaewjoho et al. 2020).
Timed Up and Go Test (TUGT) | Baseline, immediately after 6 weeks of intervention, and 1-month follow-up
  Assessing Balance Ability (TUGT) The Timed Up and Go Test (TUGT) evaluates dynamic balance and fall risk. The subject starts seated, stands up on signal, walks 3 meters around a cone, and returns to sit as quickly and safely as possible. The average time of three trials is recorded.
Static Balance Single-leg stance test (SLST) | Baseline, immediately after 6 weeks of intervention, and 1-month follow-up
  Static Balance (SLST) The Single-leg stance test assesses static balance. The subject stands on their dominant leg with the other knee bent at 90° and arms crossed over the chest. Timing measures how long the position is maintained without error (e.g., foot touching the ground, moving arms). The average time of three trials is calculated in seconds.
6-minute walk test | Baseline, immediately after 6 weeks of intervention, and 1-month follow-up
  6-Minute Walk Test (6MWT) This test assesses cardiopulmonary endurance. The subject walks as fast as possible (without running) for 6 minutes on a rectangular course (45m perimeter). Resting is allowed, but the timer continues. The total distance covered is measured to calculate VO2max.
Motor-Cognitive Dual-Task Test: | Baseline, immediately after 6 weeks of intervention, and 1-month follow-up
  Motor-Cognitive Dual-Task Test (S-TMT) The Stepping Trail Making Test assesses dual-task motor-cognitive function. The subject steps on squares numbered 1 to 16 in order as quickly and accurately as possible. The time taken to complete the sequence, including any error corrections, is recorded. The test is performed only once.
Motor-Cognitive Dual-Task Test | Baseline, immediately after 6 weeks of intervention, and 1-month follow-up
  Motor-Cognitive Dual-Task Test (F8WT) The Figure-of-8 Walk Test assesses dynamic balance and turning ability. The subject walks a figure-of-8 pattern around two cones spaced 1.5 meters apart. Time is recorded for one complete lap. In the Dual-Task variation (F8WT-MC), the subject performs the walk while holding a cup of water in their dominant hand.
Montreal Cognitive Assessment (MoCA) | Baseline, immediately after 6 weeks of intervention, and 1-month follow-up
  Assessment of Cognitive Impairment (MoCA) The MoCA test is a screening tool for cognitive impairment covering various brain functions (e.g., memory, attention). It involves a 10-15 minute interview with a maximum score of 30. A score below 26 indicates mild cognitive impairment (MCI).

CONTACTS AND LOCATIONS:
Locations (1):
- Chonticha Kaewjoho, Phayao, Thailand